CLINICAL TRIAL: NCT01417546
Title: First In-Human Phase I Trial of NHS-IL12 in Patients With Metastatic Solid Tumors
Brief Title: NHS-IL12 for Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 110225; 11-C-0225
Record Dates: First submitted 2011-08-13; First posted 2011-08-16 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Epithelial Neoplasms, Malignant; Epithelial Tumors, Malignant; Malignant Mesenchymal Tumor
Keywords: Maximum Tolerated Dose; Immune Response; Pharmacokinetics; Dose Escalation; Dose Limited Toxicity
MeSH Terms: conditions — Carcinoma; Malignant mesenchymal tumor | interventions — NHS-IL12 immunocytokine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): NHS-IL12 escalating doses on a 4 week schedule (Completed).
  Interventions: Drug: NHS-IL-12
- 2 (Experimental): NHS-IL12 escalating doses on a 2 week schedule
  Interventions: Drug: NHS-IL-12
- 3 (Experimental): NHS-IL12 expansion group on a 4 week schedule (Completed).
  Interventions: Drug: NHS-IL-12

INTERVENTIONS:
Drug: NHS-IL-12 — NHS-IL12 is an investigational agent supplied to investigators by the manufacturer EMD Serono, Inc.

SUMMARY:
Background:

- The experimental drug NHS-IL12 may help the immune system become more active and kill cancer cells that have not responded to standard treatments. NHS-IL12 has been designed to cause less severe side effects than other anticancer drugs, and may be more effective. More research is needed to test NHS-IL12 in people who have solid tumors that have not responded to treatment.

Objectives:

- To test the safety and effectiveness of NHS-IL12 as a treatment for solid tumors which have not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age with solid tumors that have not responded to standard treatments.

Design:

* Participants will be screened with a medical history, physical exam, blood and urine tests, and imaging studies.
* Participants will receive NHS-IL12 injection every 4 weeks, and will stay in the hospital for at least one day to be monitored with frequent blood tests.
* Participants will have periodic blood samples taken before treatment and during the first week after treatment for the first two cycles. They will then have blood samples taken before treatment for the rest of the cycles.

DETAILED DESCRIPTION:
Background:

* Interleukin-12 (IL-12) is a proinflammatory cytokine produced by activated phagocytes and dendritic cells (DCs) that plays a critical role in regulating the transition from innate to adaptive immunity.
* IL-12 has shown some promising clinical activity in phase I trials, including stabilization of disease in renal cancer patients with partial regression of a metastatic lesion, but has not proceeded further in clinical development due to toxicity.
* The NHS-IL12 concept is a strategy to reduce the toxicity associated with systemic administration of recombinant human IL-12 by selectively targeting delivery to tumors. The NHS-IL12 immunocytokine is composed of 2 IL-12 heterodimers, each fused to one of the H-chains of the NHS76 antibody, which has affinity for both single- and doublestranded DNA. Thus, NHS-IL12 targets delivery to regions of tumor necrosis where DNA has become exposed.

Objectives:

-To determine the dose-limiting toxicities (DLTs) and Maximum Tolerated Dose (MTD) of NHS-IL12 administered subcutaneously every 4 weeks and subcutaneously every 2 weeks in participants with metastatic or locally advanced solid epithelial or mesenchymal tumors.

Eligibility:

* Adults with histologically or cytologically proven metastatic or locally advanced solid epithelial or mesenchymal tumors, except unstable brain metastases, for which standard curative or palliative measures do not exist or are no longer effective.
* Adequate organ function as defined by liver, kidney, and hematologic laboratory testing.
* Participants with acquired immune defects, systemic autoimmune disease, history of organ transplant, history of chronic infections, or history of active inflammatory bowel disease will be excluded.

Design:

* With amendment D, this is a phase I, open-label, dose-escalation study designed to assess the safety, tolerability, PK, and biological and clinical activity of NHS-IL12. Goals are to determine the MTD of every 4-week doses at a starting dose level of 2 mcg/kg of NHS IL12 and to define the biologically optimal treatment schedule.
* Participants will be enrolled in cohorts of 3 to 6 participants using a standard 3+3 approach until MTD is reached.
* The trial will include a planned schedule-optimization amendment with up to 12 participants at each of the 2 dose levels that are of greater biologic interest (MTD and dose below MTD), which will be submitted as soon as a clear biological response (changes in circulating cytokine levels) is measured in at least 3 participants at a given dose level. With amendment L, a cohort will be enrolled evaluating NHS-IL12 at 12 mcg/kg every 2 weeks with dose escalation to 16.8 mcg/kg every 2 weeks if 0 of 3 or 1 of 6 DLTS are observed.
* With a maximum accrual ceiling of 83 participants, this study will be completed within 1year, enrolling up to 2-3 participants per month.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet the following criteria for participation:

* Participants must have histologically confirmed malignancy that is metastatic or unresectable locally advanced solid tumors.
* Participants must have completed or had disease progression on at least one prior line of disease-appropriate therapy for unresectable locally advanced or metastatic disease, or not be a candidate for therapy of proven efficacy for their disease due to an underlying physical condition.
* Participants may have disease that is measurable or non-measurable but evaluable disease (e.g. present on bone scan, rising tumor markers, non-measurable by RECIST but visible on CT scan). Participants with third space fluid (for example pleural effusions) as only site of disease will not be eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at study entry.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of NHS-IL12 in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Participants must have normal organ and marrow function as defined below:

  1. Hematological eligibility parameters (within 16 days of starting therapy):

     * Absolute granulocyte count greater than or equal to 1,500/mcL
     * Absolute lymphocyte count greater than or equal to 500/mcL
     * Platelet count greater than or equal to 100,000/mcL
     * hemoglobin greater than or equal to 9 g/dL
  2. Adequate hepatic function defined by a

     * total bilirubin level less than or equal to 1.5 times ULN or in participants with Gilbert s syndrome, a total bilirubin less than or equal to 3.0, and
     * aspartate aminotransferase (AST) and alanine-aminotransferase (ALT) levels less than or equal to 2.5 times ULN or, for participants with documented metastatic disease to the liver, AST and ALT levels less than or equal to 5 times ULN.
  3. Adequate renal function defined by an estimated creatinine clearance greater than 60 mL/min determined by 24-hour urine sampling or by the Cockcroft-Gault formula:

Ccr = (140 age) (weight, kg) (constant)/[72 times Crserum (mg/100 mL). The constant is 1 for men and 0.85 for women OR Ccr = (140 age) (weight, kg) (constant)/Crserum (micro mol/L). The constant is 1.23 for men and 1.04 for women.

CD4 lymphocyte count or other T lymphocyte subset count will not be used to determine eligibility.

* Participants must agree to practice effective contraception (both male and female subjects, if the risk of conception exists). The effects of NHS-IL12 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for 30 days after the last dose. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* A minimum of 4 weeks will be required from any prior therapy, including chemotherapy, immunotherapy and/or radiation. In addition, recovery to Grade 1 or less from reversible all reversible toxicities related to prior therapy is required at study entry. Prior immune therapy (e.g. related vaccinia and fowlpox vaccines or antigen-specific peptides) is allowed.
* Subject must sign a written informed consent document.

EXCLUSION CRITERIA:

Participants with any of the following will not be eligible for participation in this study:

* Participants who are receiving any other investigational concurrent anticancer treatment (chemotherapy, radiotherapy, immunotherapy, cytokine therapy except erythropoietin) at the time of enrollment except for disease specific appropriate hormonal therapies (e.g., ADT for prostate cancer, anti-estrogen for breast cancer, somatostatin analogue for neuroendocrine cancer)
* Concurrent use of systemic steroids (within 10 days of enrollment) will be excluded, except for physiologic doses of systemic steroid replacement or local (topical, nasal, or inhaled) steroid use. Limited doses of systemic steroids (e.g., in participants with exacerations of reactive airway disease) must have completed at least 10 days prior to enrollment. Steroid use to prevent IV contrast allergic reaction or anaphylaxis in participants who have known contrast allergies is allowed at any time prior to enrollment.
* Participants who have previously received rIL-12
* Acquired immune defects such as HIV or innate immunodeficiency because this agent requires an intact immune system. In addition, these participants are at increased risk of lethal infections when treated with marrow-altering therapy.
* Systemic autoimmune disease (e.g., lupus erythematosus, rheumatoid arthritis, Addison s disease, autoimmune disease associated with lymphoma).
* History of organ transplant.
* History of or active inflammatory bowel disease (e.g., Crohn s disease, ulcerative colitis).
* Chronic infections (e.g., hepatitis B or C, tuberculosis).
* Known hypersensitivity or allergic reactions attributed to any compounds of similar chemical or biologic composition to the study medication, such as recombinant IL-12 or other monoclonal antibodies
* Known hypersensitivity to methotrexate
* History of brain metastases because of the poor prognosis of participants with brain metastases and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke < 6 months prior to enrollment, myocardial infarction < 6 months prior to enrollment, unstable angina, congestive heart failure (greater than or equal to NYHA III) or serious cardiac arrhythmia requiring medication.
* Pulmonary disease which, in the opinion of the investigator, may impair the patient s respiratory tolerance to moderate pulmonary fluid overload (e.g., interstitial lung disease, severe chronic obstructive pulmonary disease).
* All conditions associated with significant necrosis of nontumor-bearing tissues: esophageal or gastroduodenal ulcers < 6 months prior to enrollment, organ infarction < 6 months prior to enrollment, or active ischemic bowel disease.
* Presence of medically significant third space fluid (symptomatic pericardial effusion, ascites or pleural effusion requiring repetitive paracentesis).
* History of active alcohol or drug abuse.
* Any significant disease that, in the opinion of the investigator, may impair the patient s tolerance of study treatment.
* Significant dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Pregnancy (absence to be confirmed by beta-human chorionic gonadotropin test) or lactation.
* Pleural effusion as the only evidence of metastatic disease.
* Expansion Cohorts only

  * Participants must have measurable disease, defined as at least one lesion that can be accurately measured as greater than or equal to 5 times 5 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-12-12 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) and Maximum Tolerated Dose (MTD) | During the first 6 weeks or at least 2 weeks after administration of the second dose.
  Determination of DLTs and MTD.

SECONDARY OUTCOMES:
To determine immunogenicity, safety and pharmacokinetic parameters | Ongoing
  Determination of safety, immune response and pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Portielje JE, Kruit WH, Schuler M, Beck J, Lamers CH, Stoter G, Huber C, de Boer-Dennert M, Rakhit A, Bolhuis RL, Aulitzky WE. Phase I study of subcutaneously administered recombinant human interleukin 12 in patients with advanced renal cell cancer. Clin Cancer Res. 1999 Dec;5(12):3983-9. PMID 10632329
- [Background] Mortarini R, Borri A, Tragni G, Bersani I, Vegetti C, Bajetta E, Pilotti S, Cerundolo V, Anichini A. Peripheral burst of tumor-specific cytotoxic T lymphocytes and infiltration of metastatic lesions by memory CD8+ T cells in melanoma patients receiving interleukin 12. Cancer Res. 2000 Jul 1;60(13):3559-68. PMID 10910069
- [Background] Gollob JA, Mier JW, Veenstra K, McDermott DF, Clancy D, Clancy M, Atkins MB. Phase I trial of twice-weekly intravenous interleukin 12 in patients with metastatic renal cell cancer or malignant melanoma: ability to maintain IFN-gamma induction is associated with clinical response. Clin Cancer Res. 2000 May;6(5):1678-92. PMID 10815886
- [Derived] Gatti-Mays ME, Tschernia NP, Strauss J, Madan RA, Karzai FH, Bilusic M, Redman J, Sater HA, Floudas CS, Toney NJ, Donahue RN, Jochems C, Marte JL, Francis D, McMahon S, Lamping E, Cordes L, Schlom J, Gulley JL. A Phase I Single-Arm Study of Biweekly NHS-IL12 in Patients With Metastatic Solid Tumors. Oncologist. 2023 Apr 6;28(4):364-e217. doi: 10.1093/oncolo/oyac244. PMID 36640137
- [Derived] Bekaii-Saab T, Wesolowski R, Ahn DH, Wu C, Mortazavi A, Lustberg M, Ramaswamy B, Fowler J, Wei L, Overholser J, Kaumaya PTP. Phase I Immunotherapy Trial with Two Chimeric HER-2 B-Cell Peptide Vaccines Emulsified in Montanide ISA 720VG and Nor-MDP Adjuvant in Patients with Advanced Solid Tumors. Clin Cancer Res. 2019 Jun 15;25(12):3495-3507. doi: 10.1158/1078-0432.CCR-18-3997. Epub 2019 Feb 25. PMID 30804020
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0225.html